CLINICAL TRIAL: NCT05503108
Title: DIRECT-2: Fasting Mimicking Diet Program to ImpRovE ChemoTherapy in HR+, HER2- Breast Cancer
Brief Title: Fasting Mimicking Diet Program to ImpRovE ChemoTherapy in Hormone Receptor Postive (HR+), HER2- Breast Cancer
Acronym: DIRECT-2
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: fultility
Sponsor: Leiden University Medical Center (Other)
Collaborators: The Netherlands Cancer Institute (Other); Borstkanker Onderzoek Groep (Network); Comprehensive Cancer Centre The Netherlands (Other); Koningin Wilhelmina Fonds (Other); World Cancer Research Fund International (Other); L-Nutra Inc (Industry)
Responsible Party: Principal Investigator, J.R. Kroep, Drs J.R. Kroep, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL80749.058.22 DIRECT 2; P22.028 (Other: Leiden University Medical Center (LUMC)); BOOG 2022-01 (Other: BOrstkanker Onderzoek Groep (BOOG))
Record Dates: First submitted 2022-07-24; First posted 2022-08-16 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Fasting Mimicking Diet; HER2-negative Breast Cancer; Hormone Receptor-positive Breast Cancer; Pathological Complete Response; Objective Response Rate; Neoadjuvant Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting Mimicking Diet group (Experimental): Fasting Mimicking Diet 3 days before and the day of neoadjuvant chemotherapy (ddAC, T)
  Interventions: Other: Fasting Mimicking diet program
- Normal Diet group (No Intervention): Standard neoadjuvant chemotherapy (ddAC, T)

INTERVENTIONS:
Other: Fasting Mimicking diet program — Fasting mimicking diet by L-Nutra, a 4-day low caloric, low protein, vegetarian diet 3 days prior to and the day of neoadjuvant chemotherapy administration. The FMD will take place every 4 weeks, thus in total 5 times (2x during ddAC, 3x during Paclitaxel) during the neoadjuvant chemotherapy.
  Other Names: Xentigen™
  Arms: Fasting Mimicking Diet group

SUMMARY:
In preclinical research, short-term fasting (STF) protects tumor-bearing mice against the toxic effects of chemotherapy, improves the CD8+ effector T-cell intratumor infiltration, while enhancing the chemotherapy efficacy. Short-term use of a "fasting-mimicking diet" (FMD) caused a major increase in the efficacy of cancer treatment in mice comparable to STF. In humans, the investigators recently performed a multicenter randomized phase II trial showing that patients with Human Epidermal growth factor Receptor 2 (HER2) negative breast cancer treated with neoadjuvant chemotherapy and FMD displayed a better radiological response and a better pathological response (90-100% vs <90% tumor cell reduction) than patients treated with chemotherapy without FMD (de Groot, Nat Commun 2020; NCT02126449). Therefore these findings will be validated in a phase 3 trial with the underlying hypothesis that FMD during neoadjuvant chemotherapy for breast cancer improves clinical outcomes, potentially due to improved local immunity.

DETAILED DESCRIPTION:
STF during neadjuvant chemotherapy aiming to improve the chemotherapy efficacy and decline the side effects in patients with stage II-III HR+, HER2- breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage II-III (cT1cN+ or ≥T2 any cN, cM0), HR+, HER2- breast cancer
* Detectable and measurable disease (breast and/or lymph nodes)
* World Health Organization (WHO) performance status 0-2
* Adequate organ function assessed by standard pre-treatment assessment:
* Adequate bone marrow function: white blood cells (WBCs) ≥3.0 x 109/l, neutrophils ≥1.5 x 109/l, platelets ≥100 x 109/l
* Adequate liver function: bilirubin ≤1.5 x upper limit of normal (UNL) range, ALAT and/or ASAT ≤2.5 x UNL, Alkaline Phosphatase ≤5 x UNL
* Adequate renal function: the calculated creatinine clearance should be ≥50 mL/min
* Available for treatment and follow-up
* Written informed-consent
* Willing to fill in Quality Of Life and Cognition questionnaires
* Ability to read and understand Dutch language, accessibility to a computer with internet connection and independent use of computer

Exclusion Criteria:

* Patient history of invasive or ipsilateral non-invasive breast cancer
* Active malignancy in the last 5 years, with the exclusion of basal cell carcinoma or pre-invasive cervical neoplasia/dysplasia.
* Body mass index (BMI) < 18.5 kg/m2
* Pregnancy or lactating
* Food allergy for ingredients of FMD (nuts, soy, honey)
* A metabolic condition affecting gluconeogenesis or adaptation to periodic fasting. (Diabetes Mellitus for example)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate (pCR). Both percentage of pCR and 90-100% tumor loss according to Miller & Payne | 4.5 years
Objective response rate assessed by MRI (RECIST1.1) after 4 ddAC cycles and at the end of chemotherapy | 4.5 years

SECONDARY OUTCOMES:
Determine the effect of treatment on the 3 and 5 year Event-free survival (EFS) and Overall survival (OS) | 7.5 and 9.5 years
Adverse events ≥grade 3 (maximum of total) difference between treatment arms during neoadjuvant chemotherapy (ddAC, paclitaxel and total). | 4.5 years
Quality of Life assessed by online questionnaires (EORTC QLQ-C30, EORTC QLQ-BR23), burden of therapy (Distress Thermometer) and Illness Perceptions (B-IPQ) | 5 years
  Validated online questionnaires take place at baseline, after 4 ddAC cycles, before surgery and 6 months after surgery.
Cognition assessed by Amsterdam Cognition Scan (ACS) online battery consisting of 7 online neuropsychological tests | 5 years
  online questionnaires take place at baseline, before surgery and 6 months after surgery.
Determine the effect of FMD on local immunomodulation and tumor immunity | 6 years
  By analyzing the immune-composition and gene-expression profile using multispectral Vectra imaging and Nanostring analyses respectively, in tumor samples taken at baseline (diagnostic), after 4 cycles and resection specimen

OTHER OUTCOMES:
Biomarker analysis to predict treatment outcome | 6 years
  Genetic and/or epigenetic analysis will be performed on blood samples by for example PCR and/or GWAS technique.
Optional Bioelectrical Impedance Analysis (BIA) for participants at the Leiden University Medical Center (LUMC) to investigate the change in body composition in both treatment arms. | 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Judith R Kroep, PhD, Principal Investigator — Leiden University Medical Center
Locations (7):
- Netherlands (7):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Rode Kruis ziekenhuis, Beverwijk
  - Alexander Monro Ziekenhuis, Bilthoven
  - Reinier de Graaf ziekenhuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Leiden University Medical Center, Leiden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Groot S, Lugtenberg RT, Cohen D, Welters MJP, Ehsan I, Vreeswijk MPG, Smit VTHBM, de Graaf H, Heijns JB, Portielje JEA, van de Wouw AJ, Imholz ALT, Kessels LW, Vrijaldenhoven S, Baars A, Kranenbarg EM, Carpentier MD, Putter H, van der Hoeven JJM, Nortier JWR, Longo VD, Pijl H, Kroep JR; Dutch Breast Cancer Research Group (BOOG). Fasting mimicking diet as an adjunct to neoadjuvant chemotherapy for breast cancer in the multicentre randomized phase 2 DIRECT trial. Nat Commun. 2020 Jun 23;11(1):3083. doi: 10.1038/s41467-020-16138-3. PMID 32576828
- [Background] Lugtenberg RT, de Groot S, Kaptein AA, Fischer MJ, Kranenbarg EM, Carpentier MD, Cohen D, de Graaf H, Heijns JB, Portielje JEA, van de Wouw AJ, Imholz ALT, Kessels LW, Vrijaldenhoven S, Baars A, Fiocco M, van der Hoeven JJM, Gelderblom H, Longo VD, Pijl H, Kroep JR; Dutch Breast Cancer Research Group (BOOG). Quality of life and illness perceptions in patients with breast cancer using a fasting mimicking diet as an adjunct to neoadjuvant chemotherapy in the phase 2 DIRECT (BOOG 2013-14) trial. Breast Cancer Res Treat. 2021 Feb;185(3):741-758. doi: 10.1007/s10549-020-05991-x. Epub 2020 Nov 11. PMID 33179154
- [Background] de Groot S, Pijl H, van der Hoeven JJM, Kroep JR. Effects of short-term fasting on cancer treatment. J Exp Clin Cancer Res. 2019 May 22;38(1):209. doi: 10.1186/s13046-019-1189-9. PMID 31113478
- [Background] Di Biase S, Lee C, Brandhorst S, Manes B, Buono R, Cheng CW, Cacciottolo M, Martin-Montalvo A, de Cabo R, Wei M, Morgan TE, Longo VD. Fasting-Mimicking Diet Reduces HO-1 to Promote T Cell-Mediated Tumor Cytotoxicity. Cancer Cell. 2016 Jul 11;30(1):136-146. doi: 10.1016/j.ccell.2016.06.005. PMID 27411588
- See also: Related Info — https://www.boogstudycenter.nl/studie/299/direct-2.html